CLINICAL TRIAL: NCT01608568
Title: AFFIXING POLYPROPYLENE MESH USING BARBED SUTURE (QUILL™ SRS) DURING ROBOTIC ASSISTED LAPAROSCOPIC SACROCOLPOPEXY RANDOMIZED CONTROLLED TRIAL
Brief Title: Affixing Polypropylene Mesh Using Barbed Suture (Quill™ SRS) During Robotic Assisted Laparoscopic Sacrocolpopexy
Acronym: Quill RALSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jasmine Tan-Kim, Urogynecologist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Robotic Sacrocolpopexy Quill
Record Dates: First submitted 2012-02-29; First posted 2012-05-31 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Prolapse
Keywords: Sutures; Pelvic Organ Prolapse; Sacrocolpopexy; Robotic Assisted Laparoscopy
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrupted suture (Active Comparator): interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA)
  Interventions: Device: Device is the type of suture used: Quill suture vs. Interrupted suture
- Quill suture (Active Comparator): self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada)
  Interventions: Device: Device is the type of suture used: Quill suture vs. Interrupted suture

INTERVENTIONS:
Device: Device is the type of suture used: Quill suture vs. Interrupted suture — To compare two methods of polypropylene mesh attachment during robotic assisted laparoscopic sacrocolpopexy (RALSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).
  Other Names: (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) (PDS II™, Ethicon, Somerville, NJ, USA)

SUMMARY:
1.0 STUDY OBJECTIVE 1.1 PRIMARY OBJECTIVE - To compare two methods of polypropylene mesh attachment during robotic assisted laparoscopic sacrocolpopexy (RALSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

1.2 SECONDARY OBJECTIVE - To compare robotic assisted laparoscopic sacrocolpopexy anatomic failure rates at 6 months post-operative follow-up using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA). The investigators will also assess mesh erosion rates, costs, and surgeon satisfaction rates.

2.0 HYPOTHESIS 2.1 Primary: 2.1.a. Attachment of mesh using the running technique with self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) will be faster than the standard fixation interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

2.2 Secondary: 2.2.a. Attachment of mesh using the running technique with self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) will be less costly than the standard fixation interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

2.2.b. Failure rates and mesh erosion rates for each technique will be equally low.

2.2.c. Surgeons will prefer the barbed running technique over the interrupted technique based on subjective surgeon satisfaction questionnaires.

ELIGIBILITY:
INCLUSION CRITERIA

* >18 years old
* Undergoing RALSC with or without other procedures for pelvic organ prolapse or incontinence
* Willing to return for follow-up visits
* Written informed consent obtained from each subject
* Must be having a robotic assisted laparoscopic sacrocolpopexy

Exclusion Criteria:

* Decline to participate
* Pregnant or contemplating future pregnancy
* Unable to participate in the informed consent process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Mesh attachment interval | Intraoperative placement of mesh - approximately 30 minutes to 2 hours
  To compare two methods of polypropylene mesh attachment during robotic assisted laparoscopic sacrocolpopexy (RALSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA)in terms of time.

SECONDARY OUTCOMES:
Anatomic outcomes using the two suture types | 6 months post-operatively
  To compare robotic assisted laparoscopic sacrocolpopexy anatomic failure rates at 6 months post-operative follow-up using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA). We will also assess mesh erosion rates, costs, and surgeon satisfaction rates.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Tan-Kim J, Nager CW, Grimes CL, Luber KM, Lukacz ES, Brown HW, Ferrante KL, Dyer KY, Kirby AC, Menefee SA. A randomized trial of vaginal mesh attachment techniques for minimally invasive sacrocolpopexy. Int Urogynecol J. 2015 May;26(5):649-56. doi: 10.1007/s00192-014-2566-8. Epub 2014 Nov 25. PMID 25421934